CLINICAL TRIAL: NCT03408054
Title: The Relaxant Effect of Nitroglycerin on Oxytocin Desensitized Human Myometrium and the Return of Contractility on Re-exposure to Oxytocin- an in Vitro Study
Brief Title: The Relaxant Effect of Nitroglycerin on Oxytocin Desensitized Human Myometrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Oxytocin; Nitroglycerin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): No oxytocin desensitization (pretreatment), no nitroglycerin
- Oxytocin desensitized - no nitroglycerin (Active Comparator): Pretreated with oxytocin, no nitroglycerin exposure
  Interventions: Drug: Oxytocin
- Oxytocin desensitized - plus nitroglycerin (Active Comparator): Pretreated with oxytocin followed by nitroglycerin exposure
  Interventions: Drug: Oxytocin; Drug: Nitroglycerin
- Non oxytocin desensitized - plus nitroglycerin (Active Comparator): No oxytocin pretreatment, followed by nitroglycerin exposure
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 10-5M solution
  Other Names: Duratocin, pitocin
  Arms: Oxytocin desensitized - no nitroglycerin; Oxytocin desensitized - plus nitroglycerin
Drug: Nitroglycerin — Nitroglycerin 25-1000mcg
  Arms: Non oxytocin desensitized - plus nitroglycerin; Oxytocin desensitized - plus nitroglycerin

SUMMARY:
Oxytocin causes myometrial contraction via the oxytocin receptor (OTR). Desensitization of the OTR after exposure to oxytocin has been demonstrated in previous studies. The resultant need for a higher oxytocin dose to cause adequate uterine contraction in vivo has also been demonstrated in laboring women having received oxytocin for labor augmentation.

Achieving rapid uterine relaxation can be invaluable for maternal and fetal wellbeing in some acute obstetric emergency settings. Nitroglycerin has become a commonly used agent for achieving rapid uterine relaxation amongst obstetric anesthesiologists.

Previous studies have concluded that oxytocin can be used to re-establish uterine tone following nitroglycerin mediated relaxation. However, no studies to date have looked at the effects of nitroglycerin mediated relaxation of uterine muscle that has undergone oxytocin receptor desensitization. Nor has the response to oxytocin re-exposure and return of contractility in desensitized myometrium (following nitroglycerin) been examined.

The investigators hypothesize that nitroglycerin will reduce and inhibit uterine contractions in both oxytocin pre-treated myometrium, as well as untreated myometrium in a dose dependent fashion, but that myometrium that has undergone OTR desensitization will require less nitroglycerin for contractions to abate.

The investigators also expect that the dose of oxytocin required to re-establish equivalent contractions will be higher in the myometrial samples which have undergone nitroglycerin mediated relaxation.

DETAILED DESCRIPTION:
Oxytocin and nitroglycerin have opposing actions on the myometrium. The pharmacological properties of quick onset and offset of action of nitroglycerin have made this the preferred drug to be used in acute scenarios where uterine relaxation is necessary.

As nitroglycerin causes changes to intracellular calcium levels and the ability uterine muscle to engage in effective contraction, it is plausible that the effects of nitroglycerin may interfere with subsequent uterine contractility and action of oxytocin.

The situation where a difficult fetal extraction is encountered at cesarean section may be in two broad groups of patients. Those pre-exposed to oxytocin and those with an oxytocin naïve myometrium. Given the large observational variation in dosages of nitroglycerin usage seen in the literature we feel it is vital to investigate whether pre-exposure to oxytocin impacts on the ability of nitroglycerin to relax uterine smooth muscle. Furthermore, once the uterus has relaxed following nitroglycerin exposure, is there a need for higher doses of oxytocin to be administered in order to re-engage the uterus in effective contraction? And is this requirement further exacerbated by the phenomenon of oxytocin receptor desensitization? These clinically important questions will be addressed by the design of this in vitro myometrial study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean delivery or first repeat Cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous Cesarean delivery
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency Cesarean section in labor
* Patients with medical/pregnancy related conditions, such as diabetes, preeclampsia and essential hypertension

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Motility Index | 8 hours
  Motility index (MI) takes into account both the amplitude and frequency of the myometrial contraction. It is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 8 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 8 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jayasooriya GS, Carvalho JCA, Luca A, Balki M. The Effects of Nitroglycerin on the Oxytocin Dose-Response Profile in Oxytocin-Desensitized and Naive Human Myometrium: An In Vitro Study. Anesth Analg. 2021 Jan;132(1):231-239. doi: 10.1213/ANE.0000000000005055. PMID 32858531